CLINICAL TRIAL: NCT01906138
Title: A Prospective, Open Label Study Assessing the 24-hour Intraocular Pressure Pattern Monitored by SENSIMED Triggerfish® in Primary Angle Closure and Primary Angle Closure Glaucoma Patients, Before and After Laser Peripheral Iridotomy
Brief Title: An Open Label Study Assessing the 24-hour Intraocular Pressure Pattern in PAC and PACG Patients, Before and After Laser Peripheral Iridotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1106
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENSIMED Triggerfish® (Other): All eligible patients will be assigned to 24-hour intraocular pressure recording using Triggerfish
  Interventions: Device: SENSIMED Triggerfish®

INTERVENTIONS:
Device: SENSIMED Triggerfish® — All eligible patients will be assigned to 24-hour intraocular pressure recording using Triggerfish

SUMMARY:
The purpose of the study is to determine the relationship of the intraocular pressure patterns recorded during 2 sessions using Triggerfish, before and after elective laser peripheral iridotomy in angle closure glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary angle closure (PAC) or primary angle closure glaucoma (PACG) with indication for laser peripheral iridotomy (PAC is defined by the presence of a partial or complete iridotrabecular contact in more than 2 quadrants with either raised intraocular pressure [i.e. more than 21 mmHg] and/or primary adhesion to the trabecular meshwork (peripheral anterior synechiae [PAS]; however, with normal optic disc and visual field. PACG is defined by the presence of iridotrabecular contact with either raised intraocular pressure and/or PAS, and evidence of glaucomatous optic disc and visual field)
* No intraocular pressure-lowering drug treatment or a 4-week wash-out period prior to study day 0 and throughout the study
* Aged ≥18 years, of either sex
* Not more than 6 diopters spherical equivalent on the study eye
* Not more than 2 diopters cylinder equivalent on the study eye
* Have given written informed consent, prior to any investigational procedure

Exclusion Criteria:

* History of acute angle closure glaucoma
* Secondary angle closure glaucoma
* History of ocular surgery within the last 3 months
* History of ocular laser treatment, including previous laser peripheral iridotomy
* Corneal or conjunctival abnormality precluding contact lens adaptation
* Severe dry eye syndrome
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The 24-hour Intraocular pressure pattern as recorded by Triggerfish in patients with Primary Angle Closure and Primary Angle Closure Glaucoma | 24 hours

SECONDARY OUTCOMES:
To assess the nycthemeral Intraocular pressure patterns specific to PAC and PACG | 24 hours
To assess the effect of laser peripheral iridotomy on diurnal and nocturnal intraocular pressure pattern for each group of patients | 24 hours
To assess the comfort of contact lens sensor wear in patients of Indian origin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shibal Bhartiya, MD, Principal Investigator — Fortis Memorial Research Institute
Locations (1):
- Fortis Memorial Research Institute, Glaucoma facility, Haryāna, Haryana, India